CLINICAL TRIAL: NCT04426604
Title: Validity of Fluorescence-Based Devices Versus Visual-Tactile Method in Detection of Secondary Caries Around Resin Composite Restorations: Invivo Diagnostic Accuracy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Adly, Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AMAI-CU-2020-06-07
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Secondary Caries Around Resin Composite Restorations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be blind about the type of intervention/control assessment methods. However it will not be allowed amongst the examiners to exchange any information throughout the entire study period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light induced fluorescence intraoral camera (Experimental)
  Interventions: Diagnostic Test: Light induced fluorescence intraoral camera
- Laser-induced fluorescence device (Experimental)
  Interventions: Diagnostic Test: Laser-induced fluorescence device
- Visual-tactile assessment method according to FDI criteria (Active Comparator)
  Interventions: Diagnostic Test: Visual-tactile assessment method according to FDI criteria

INTERVENTIONS:
Diagnostic Test: Light induced fluorescence intraoral camera — Each restoration margins will be assessed by Light induced fluorescence intraoral camera to assess its validity in diagnosing secondary caries around margins of resin composite restorations
  Arms: Light induced fluorescence intraoral camera
Diagnostic Test: Laser-induced fluorescence device — Each restoration margins will be assessed by Laser-induced fluorescence device to assess its validity in diagnosing secondary caries around margins of resin composite restorations
  Arms: Laser-induced fluorescence device
Diagnostic Test: Visual-tactile assessment method according to FDI criteria — Each restoration margins will be assessed by visual-tactile assessment method which includes the use of mirror, probe under good illumination condition to assess its validity in diagnosing secondary caries around margins of resin composite restorations
  Arms: Visual-tactile assessment method according to FDI criteria

SUMMARY:
This study will be conducted to evaluate the clinical performance and validity of both light-induced fluorescence intraoral camera and laser-induced fluorescence device in comparison to visual-tactile assessment method in detection of secondary caries around margins of resin composite restorations.

DETAILED DESCRIPTION:
Each patient should have at least one resin composite restoration. The restoration will be evaluated by all diagnostic methods. Each examiner will independently record the dental findings using all methods, the visual- tactile assessment method and both fluorescent-aided identification methods. The visual-tactile assessment method includes the use of mirror, probe under good illumination condition, while the fluorescent-aided identification methods will be performed by both light-induced fluorescence intraoral camera and laser-induced fluorescence device. Then Diagnostic performance for caries detection was evaluated, assessing the validity of each diagnostic method in diagnosing secondary caries around margins of resin composite restorations

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 years of age.
* Patients should have an acceptable oral hygiene level.
* Patients should have at least one resin composite restoration.

Exclusion Criteria:

* Patients with a compromised medical history.
* Patients with active severe periodontal disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Validity of Fluorescence-based Devices versus Visual-tactile method | Through study completion, an average of 5 months
  Diagnostic performance for caries detection was evaluated, assessing the validity of each diagnostic method in diagnosing secondary caries around margins of resin composite restorations in terms of sensitivity and specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Adly AM, Ibrahim SH, El-Zoghbi AF. Clinical validity of fluorescence-based devices versus visual-tactile method in detection of secondary caries around resin composite restorations: diagnostic accuracy study. BDJ Open. 2025 Jan 6;11(1):2. doi: 10.1038/s41405-024-00284-7. PMID 39762230